CLINICAL TRIAL: NCT04016909
Title: The Effect of Combined Aerobic Exercise and Calorie Restriction on Mood, Cognition, and Motor Behavior in Overweight and Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LithuanianSportsU-1
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: brain activity; cognitive function; diet; exercise; motor behavior; psychosocial state
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise plus calorie restriction (Experimental): The experimental intervention: both exercise and calorie restriction, as described below:
  Exercise intervention. 6 months, 72 supervised aerobic exercise training sessions on cycle ergometers, including 3 sessions of training per week. A warm-up procedure consisting of 5 min of low-intensity stretching was completed by all women before the aerobic training. Subsequently, a 50 min aerobic training at an intensity between 60% and 70% of the maximum heart rate (HR) was performed. Thereafter, a cool-down consisting of 5 min of low-intensity stretching and breathing exercises was completed. HR was recorded continuously throughout the training sessions using an HR monitor (S625X, Polar Electro, Kempele, Finland).
  Calorie restriction intervention. The CR intervention was designed to create a 12.5% energy deficit, with the goal of reducing body weight by 5%-10% over 6 months.
  Interventions: Procedure: aerobic exercise plus calorie restriction
- Control (No Intervention): No intervention and participants were instructed to maintain their regular physical activity and diet regime for 6 months; they were also prohibited from participating in any weight-loss or exercise program.

INTERVENTIONS:
Procedure: aerobic exercise plus calorie restriction — both a 6-month aerobic exercise program (moderate intensity) and caloric restriction (12.5% energy deficit)
  Arms: aerobic exercise plus calorie restriction

SUMMARY:
The benefits of weight-loss programs on mood state and cognitive and motor behavior remain unclear and are largely limited to those of calorie restriction (CR) or physical exercise alone. Our aim was to investigate the effect of a combined CR and aerobic exercise program on mood state, cognition-related brain activity, and cognitive and motor behavior in overweight and obese women. Twenty-six overweight or obese women were randomized to either a control group (no intervention) or an experimental group (aerobic exercise + 12.5% energy-intake reduction). Brain-derived neurotrophic factor (BDNF) levels, mood, prefrontal cortex activity, cognitive performance, and learning of a speed-accuracy task were evaluated before and 6 months after the beginning of the program. Confusion and depression increased in the control group (P < 0.05), whereas tension decreased in the experimental group (P < 0.05). BDNF level and learning of a speed-accuracy task remained unchanged. Although PFC activity and executive functions were not affected, the reaction time of visual scanning and associative learning were improved in the experimental group (P < 0.05). An improvement in reaction time during the speed-accuracy task was observed (P < 0.05). In conclusion, a 6-month combined CR and aerobic exercise intervention improved the psychosocial mental state of overweight and obese women. Although it improved motor planning during the speed-accuracy task, it had little impact on cognition and no effect on brain activity and learning of the speed-accuracy task.

ELIGIBILITY:
Inclusion Criteria:

* gender: female;
* body mass index (BMI) greater than 25 kg/m2;
* exhibiting weight stability (body weight change <2 kg) for at least 2 months prior to enrollment;
* sedentary lifestyle (regular exercise 1 h/week).

Exclusion Criteria:

* undergoing lactation;
* pregnant or postmenopausal;
* type 2 diabetes;
* cardiovascular disease.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Weight | baseline
  weight (TBF-300 body composition scale; Tanita, UK Ltd., UK) was measured while the participants wore only underwear and were barefoot.
mood state | baseline
  Mood was assessed using the 24-item Brunel Mood Scale, which estimates anger, confusion, depression, fatigue, tension, and vigor. Items are rated on a 5-point Likert scale anchored by 0 (not at all) and 4 (extremely), according to how participants feel "right now."
Blood brain-derived neurotrophic factor (BDNF) | baseline
  Venous blood samples (5 mL) were collected and allowed to clot at room temperature. Serum was then separated by centrifugation for 15 min at 1,200 g (room temperature) and stored at -80°C until analysis. BDNF were measured using an enzyme-linked immunoassay system (Gemini; Stratec Biomedical, Birkenfeld, Germany).
Height | baseline
  Body height was measured in meters with an accuracy of 5 mm
Cognitive functions | baseline
  Automated Neuropsychological Assessment Metrics Version 4 (ANAM-4; Vista Life, USA) was used to measure neurocognitive skills: motor reaction time, mental flexibility, mathematical processing, working memory, visual scanning and associative learning skills. Participants were familiarized with the test battery twice before the experiments.
prefrontal cortex activity | baseline
  Assessment of brain activity was performed on a continuous wave system (fNIR Imager 1100, fNIR Devices LLC, Potomac, MA, United States) using a flexible 16 optode probe set. The sensor has a temporal resolution of 500 ms per scan with a 2.5 cm source-detector separation allowing for approximately 1.25 cm penetration depth and 16 measurement locations on a rectangular grid covering the forehead region, designed to observe dorsal and inferior frontal cortical areas.
psychomotor function | baseline
  During the speed-accuracy task, the participant was required to position the handle symbol (0.0035 m in diameter) in the start zone on the computer screen. The participant then had to react to the target (a green circle, 0.007 m in diameter) on the computer screen as fast as possible and to push the handle of the device so that the circle of the handle symbol reached the target as quickly and accurately as possible. The distance from the start zone to the target was 0.17 m. The endpoint of the movement was reached when the center of the handle symbol stopped in the circle and stayed there for at least 0.02 s.

SECONDARY OUTCOMES:
Changes in body weight | 6 months
  weight (TBF-300 body composition scale; Tanita, UK Ltd., UK) was measured while the participants wore only underwear and were barefoot.
Changes in mood state | 6 months
  Mood was assessed using the 24-item Brunel Mood Scale, which estimates anger, confusion, depression, fatigue, tension, and vigor. Items are rated on a 5-point Likert scale anchored by 0 (not at all) and 4 (extremely), according to how participants feel "right now."
changes in blood brain-derived neurotrophic factor (BDNF) | 6 months
  Venous blood samples (5 mL) were collected and allowed to clot at room temperature. Serum was then separated by centrifugation for 15 min at 1,200 g (room temperature) and stored at -80°C until analysis. BDNF were measured using an enzyme-linked immunoassay system (Gemini; Stratec Biomedical, Birkenfeld, Germany).
Improvement of cognitive functions | 6 months
  Automated Neuropsychological Assessment Metrics Version 4 (ANAM-4; Vista Life, USA) was used to measure neurocognitive skills: motor reaction time, mental flexibility, mathematical processing, working memory, visual scanning and associative learning skills. Participants were familiarized with the test battery twice before the experiments.
Changes in prefrontal cortex activity | 6 months
  Assessment of brain activity was performed on a continuous wave system (fNIR Imager 1100, fNIR Devices LLC, Potomac, MA, United States) using a flexible 16 optode probe set. The sensor has a temporal resolution of 500 ms per scan with a 2.5 cm source-detector separation allowing for approximately 1.25 cm penetration depth and 16 measurement locations on a rectangular grid covering the forehead region, designed to observe dorsal and inferior frontal cortical areas.
Improvement of psychomotor function | 6 months
  During the speed-accuracy task, the participant was required to position the handle symbol (0.0035 m in diameter) in the start zone on the computer screen. The participant then had to react to the target (a green circle, 0.007 m in diameter) on the computer screen as fast as possible and to push the handle of the device so that the circle of the handle symbol reached the target as quickly and accurately as possible. The distance from the start zone to the target was 0.17 m. The endpoint of the movement was reached when the center of the handle symbol stopped in the circle and stayed there for at least 0.02 s.

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Zlibinaite, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No